CLINICAL TRIAL: NCT02301247
Title: Treating New Learning and Memory Deficits in Progressive Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: International Progressive MS Alliance (Unknown)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuroscience and Neuropsychology Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-839-14
Record Dates: First submitted 2014-11-17; First posted 2014-11-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis, Progressive; Cognition - Other; Memory Impairment
Keywords: Multiple Sclerosis, Progressive; cognition; memory; treatment
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive memory retraining exercises administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Memory retraining exercises
- Placebo (Placebo Comparator): The placebo group will receive placebo control memory exercises administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Placebo control memory exercises

INTERVENTIONS:
Behavioral: Memory retraining exercises — Memory retraining exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Arms: Experimental Group
Behavioral: Placebo control memory exercises — Placebo control memory exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Arms: Placebo

SUMMARY:
This study is a double-blind placebo-controlled randomized clinical trial (RCT) to provide Class I evidence in support of or in refute of the efficacy of the modified Story Memory Technique (mSMT) in persons with progressive MS, with outcome measured through three mechanisms: (1) a traditional neuropsychological evaluation (NPE) (2) an assessment of global functioning (AGF) examining the impact of the treatment on daily activities, and (3) an optional functional magnetic resonance imaging (fMRI) scan.

DETAILED DESCRIPTION:
There is a clear unmet need in the clinical care of persons with Progressive MS - there are no treatments for memory dysfunction with demonstrated efficacy in persons with progressive disease. This is despite the fact that cognitive impairment is a major contributor to unemployment and decreased functional status in MS and memory deficits are a major source of such disability. The investigator recent RCT's demonstrated the modified Story Memory Technique (mSMT) to be effective for improving new learning and memory in individuals with MS, demonstrating efficacy across three realms of functioning, objective behavior, brain functioning and everyday life. This convincing data provides Class I evidence supporting the efficacy of the mSMT for improving new learning and memory in MS. However, treatment efficacy was not adequately tested in the progressive MS population. This is a major limitation due to the fact that progressive MS carries with it major cognitive difficulties, of which learning and memory are one of the most common. The currently proposed RCT will address this limitation. The investigators will use methodologically vigorous research design to provide Class I evidence in support of or in refute of the efficacy of the mSMT in persons with progressive MS, with outcome measured through three mechanisms: (1) a traditional neuropsychological evaluation (NPE) (2) an assessment of global functioning (AGF) examining the impact of the treatment on daily activities and (3) an optional functional magnetic resonance imaging (fMRI) scan. Both groups will undergo baseline, immediate follow-up, and 3-month follow-up assessments

Thus, the current study will objectively evaluate the clinical utility of the mSMT to improve new learning and memory in individuals with progressive MS with documented deficits in this area. This protocol has been previously utilized in a Relapsing-Remitting MS sample, yielding exceptional outcome data. Pilot data in a small sample of progressive MS patients is promising. The investigators will also increase the generalizability and real life application of assessment techniques by assessing outcome following cognitive retraining with more global measures of everyday life. Finally, the long-term efficacy of the mSMT will be evaluated in progressive MS through the inclusion of a 3-month follow-up assessment. Given the absence of any treatment for impaired learning and memory in progressive patients, the results of the present RCT will have a significant impact on symptom management and quality of life for persons with Progressive MS.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 30 and 59
* diagnosed with Progressive Multiple Sclerosis
* have visual acuity of better then 20/60 in worse eye

Exclusion Criteria:

* has a prior stroke or neurological injury/disease (brain tumor, epilepsy, traumatic brain injury).
* has a history of psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis).
* currently taking medications such as: steroids, benzodiazepines, and neuroleptics. .
* difficulty with vision, eyesight worse then 20/60, or has diminished sight in visual field, double vision, or nystagmus.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2017-04-02 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
Change in scores on standardized neuropsychological tests of memory | Scores will be assessed at three time-points: Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention

SECONDARY OUTCOMES:
Change in scores on self-report of emotional functioning, measured via questionnaire | Scores will be assessed at three time-points: Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention
Change in scores on self-report of memory functioning, measured via questionnaire | Scores will be assessed at three time-points: Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention
Change in scores on self-report of quality of life, measured via questionnaire | Scores will be assessed at three time-points: Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Weiner, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States